CLINICAL TRIAL: NCT01791634
Title: Prospective, Randomized, Multi-Center Clinical Evaluation of the Open Wedge Osteotomy and Low Profile Plate & Screw (LPS) System Compared to the Proximal Chevron Osteotomy for the Treatment of Hallux Valgus With an Increased Intermetatarsal Angle
Brief Title: Prospective, Multi-Center Clinical Evaluation of the Open Wedge Osteotomy and Low Profile Plate & Screw (LPS) System Compared to the Proximal Chevron Osteotomy for the Treatment of Hallux Valgus With an Increased Intermetatarsal Angle
Acronym: Hallux valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Glazebrook, Associate Professor,Dalhousie University Orthopedics, Nova Scotia Health Authority
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version1 Jan 4 2007
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- proximal open wedge osteotomy with LPS system (Experimental): Proximal open wedge osteotomy with Low profile plate and screws
  Interventions: Procedure: proximal open wedge osteotomy with LPS system
- proximal wedge osteotomy (Active Comparator): Proximal wedge osteotomy procedure
  Interventions: Procedure: proximal chevron osteotomy

INTERVENTIONS:
Procedure: proximal chevron osteotomy
  Arms: proximal wedge osteotomy
Procedure: proximal open wedge osteotomy with LPS system
  Arms: proximal open wedge osteotomy with LPS system

SUMMARY:
Is there a difference in clinical outcome measures as assessed by the AOFAS, SF-36 and Visual Analogue Scale of adult patients with moderate to severe hallux valgus with increased intermetatarsal angles treated with a proximal open wedge osteotomy with LPS system versus the proximal chevron osteotomy?

DETAILED DESCRIPTION:
Is there a difference in radiologic outcomes of adult patients with moderate to severe hallux valgus with increased intermetatarsal angles treated with a proximal open wedge osteotomy with LPS system versus proximal wedge osteotomy? Is there a difference in surgical times or surgeon procedure preference in the treatment of adult patients with moderate to severe hallux valgus with increased intermetatarsal angles treated with a proximal open wedge osteotomy with LPS system versus proximal wedge osteotomy? Is there a difference in complication rates of adult patients with moderate to severe hallux valgus with increased intermetatarsal angles treated with a proximal open wedge osteotomy with LPS system versus proximal wedge osteotomy?

ELIGIBILITY:
Inclusion Criteria:

* age (> 16 years of age) moderate to severe hallux valgus angle [HVA] of >30º with increased intermetatarsal angles [IMA] of >13º
* persistent incapacitating symptoms despite non-operative treatment (shoe wear modification, orthoses, non-steroidal anti-inflammatory drugs and restricted activity)

Exclusion Criteria:

* degenerative arthritis of 1st metatarsophalangeal (MTP) joint
* neuropathic patients
* diabetes mellitus
* peripheral vascular disease
* previous 1st metatarsal, hallux or MTP joint surgery
* active or recent foot/toe infection
* currently participation in a another clinical trial
* Worker's Compensation Board patients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Short Form 36 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mark A Glazebrook, MSc PhD Dip Sports Med MD,FRCS, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada